CLINICAL TRIAL: NCT05123651
Title: A Randomized, Double-blinded, Parallel, Placebo-controlled Study to Investigate the Efficacy of Lb Rhamnosus [Junlebao Lr. X253] as Oral Probiotics
Brief Title: Research on the Characteristics and Application of Lactobacillus Rhamnosus X253 as Oral Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Junlebao Dairy Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: L.r X253 as oral probiotics
Record Dates: First submitted 2021-10-18; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: A total of 60 volunteers were recruited and randomly divided into three groups with 20 people in each group. Among them, 17 volunteers terminated the experiment due to taking antibiotics and hormone drugs during the experiment. The remaining 43 volunteers belonged to three different groups: Control group (n=16), Viable group (n=13), Inactivated group (n=14).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): who met inclusion criteria, will receive an identical X253 Probiotic lozenge Supplement looking and tasting placebo.
  Interventions: Biological: Lactobacillus rhamnosus X253
- Viable group (Experimental): who met inclusion criteria, will receive an identical X253 Probiotic lozenge(containing active L.r X253).
  Interventions: Biological: Lactobacillus rhamnosus X253
- Inactivated group (Experimental): who met inclusion criteria, will receive an identical X253 Probiotic lozenge(containing inactive L.r X253).
  Interventions: Biological: Lactobacillus rhamnosus X253

INTERVENTIONS:
Biological: Lactobacillus rhamnosus X253 — Every two weeks, all volunteers were given the number of probiotic lozenges to be used within two weeks. Edible method: 3 times a day, 1 tablet every time (0.8g/tablet). Put the tablet in the mouth and keep it in the mouth for at least 2-3 minutes before swallowing. Take it once every 30 minutes after breakfast, lunch and dinner. Do not brush your teeth, eat foods, or rinse your mouth within half an hour of consumption. Maintain oral hygiene according to the original habits during consumption, and do not use fluoride toothpaste during consumption.

SUMMARY:
The aim of the study is to study the application of Lactobacillus rhamnosus X253 as oral probiotics by the way of a randomised, double blinded, parallel, placebo-controlled clinical trial, and to eto detect the changes in oral flora of volunteers, and judge the improvement effect of X253 lozenges on the human oral flora.

DETAILED DESCRIPTION:
population experiments were carried out, and Quantitative Real-time PCR was used to detect the expression level of the target strains in volunteers' oral, High-throughput sequencing technology to detect the changes in oral flora of volunteers, and judge the improvement effect of X253 lozenges on the human oral flora. The effects of X253 lozenges on the volunteers' oral odor, defecation frequency and gum bleeding was surveyed and conuted by questionnaire.

ELIGIBILITY:
1. Age: 18 years old and above;
2. Gender: There is no restriction on men or women (women are not pregnant);
3. Keep more than 20 original teeth in the oral cavity;
4. Have not had periodontal treatment, tooth whitening (ceramic veneer, cold light whitening), orthodontics, etc. in the past 6 months;
5. No oral topical medication (such as mouthwash, watermelon frost) within 1 month;
6. No dental filling plan in the next 2-6 weeks;
7. Have not taken antibiotics (such as amoxicillin, cephalosporin, roxithromycin, ofloxacin, etc.), hormones (such as glucocorticoids, thyroid hormones, insulin, etc.) and immunosuppressive agents(such as dexamethasone, methylprednisolone, sirolimus, azathioprine) in the past half month; no taking plan for antibiotics (such as amoxicillin, cephalosporin, roxithromycin, ofloxacin, etc.), hormones (such as glucocorticoids, thyroid hormones, insulin, etc.) and immunosuppressive agents (such as dexamethasone, methylprednisolone, sirolimus, azathioprine) within the next 2-6 weeks;
8. No obvious abnormal occlusal relationship (the corresponding relationship between the upper jaw and the lower jaw is not normal, and the chewing efficiency is low).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-14 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Porphyromonas gingivalis(P.g), Streptococcus mutans(S.m), Streptococcus gordonii(S.g), and Bifidobacterium(Bif) gene expression from tartar samples | week 2 during the intervention
  In a sterile operating table, place the collected dental floss in a 180μL lysozyme (20mg/mL) water bath, use a DNA extraction kit (Tiangen Biotechnology Co., Ltd.) to extract the DNA in the oral sample, and store the DNA sample at -20°C. Quantitative Real-time PCR (Tiangen Biotechnology Co., Ltd.) was performed for the Porphyromonas gingivalis(P.g), Streptococcus mutans(S.m), Streptococcus gordonii(S.g), and Bifidobacterium(Bif) contained in the DNA of the tartar sample. The experiment results at 0 weeks were used as the control, and the relative quantitative method which is named 2-∆∆ct method was used to calculate the gene expression level of the target bacteria in the 2th week.
Porphyromonas gingivalis(P.g), Streptococcus mutans(S.m), Streptococcus gordonii(S.g), and Bifidobacterium(Bif) gene expression from tartar samples | week 4 during the intervention
  In a sterile operating table, place the collected dental floss in a 180μL lysozyme (20mg/mL) water bath, use a DNA extraction kit (Tiangen Biotechnology Co., Ltd.) to extract the DNA in the oral sample, and store the DNA sample at -20°C. Quantitative Real-time PCR (Tiangen Biotechnology Co., Ltd.) was performed for the Porphyromonas gingivalis(P.g), Streptococcus mutans(S.m), Streptococcus gordonii(S.g), and Bifidobacterium(Bif) contained in the DNA of the tartar sample. The experiment results at 0 weeks were used as the control, and the relative quantitative method which is named 2-∆∆ct method was used to calculate the gene expression level of the target bacteria in the 4th week.

SECONDARY OUTCOMES:
changes of oral problems | 1 week during the intervention
  Design a questionnaire about the improvement of oral problems, and distribute it to the volunteers every week, then collect and organize the data.

CONTACTS AND LOCATIONS:
Locations (1):
- Shijiazhuang JunlebaoDairy Co.Ltd., Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided